CLINICAL TRIAL: NCT00067990
Title: Angiotensin II Blockade for the Prevention of Cortical Interstitial Expansion and Graft Loss in Kidney Transplant Recipients
Brief Title: Angiotensin II Blockade for Chronic Allograft Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ANGIOB; R01DK060706 (NIH); NCT01467895 (obsolete NCT alias)
Record Dates: First submitted 2003-09-03; First posted 2003-09-05 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Kidney Disease; Proteinuria
Keywords: chronic allograft nephropathy; post transplant proteinuria
MeSH Terms: conditions — Kidney Diseases; Proteinuria | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Losartan 100mg (Experimental): Losartan 100 mg per day to be started within three months of transplantation and continuing treatment for five years.
  Interventions: Drug: Losartan 100mg
- Placebo (Placebo Comparator): No intervention with continuing follow-up for five years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan 100mg — To be started within three months of transplant and continued for five years.
  Other Names: Losartan
  Arms: Losartan 100mg
Drug: Placebo — No treatment with continued follow-up for five years.
  Arms: Placebo

SUMMARY:
Chronic allograft nephropathy continues to be a major cause of kidney transplant loss and return to dialysis. Treatment options are limited and the course of the disease tends to be progressive. This trial is designed to prevent a major mediator of this process, namely the expansion of the cortical interstitial compartment of the kidney where most of the scarring occurs. The drug being studied, Losartan, has proven efficacious in a number of kidney diseases.

DETAILED DESCRIPTION:
Renal transplant loss due to chronic allograft nephropathy (CAN) is widely acknowledged as a major problem that has increased in relative importance as the incidence of early graft loss from acute rejection has declined. Studies from various centers, including the University of Minnesota, suggest that, after excluding patients dying with a functioning graft, as many as 80% of patients who will return to dialysis do so because of CAN. At the present time there are no therapeutic options once the clinical manifestations of CAN have developed. Testing measures to prevent CAN have not been addressed.

The overall purpose of this project is to investigate the role of the renin-angiotensin-aldosterone system (RAAS) in the development of CAN. This system plays an important role in the progression of many experimental and clinical renal diseases. Furthermore, blockade of this system with angiotensin converting enzyme inhibitors and angiotensin II receptor blockers has yielded beneficial results in retarding injury and progression in numerous intrinsic renal diseases. This study specifically investigates the long term benefit of the angiotensin II receptor blocker, losartan, in the prevention of cortical interstitial volume expansion (an accurate predictor of long term graft function) and graft loss from biopsy proven CAN in a 5 year, randomized, double masked, placebo controlled study of kidney transplant recipients. This clinical trial will directly test the hypothesis that blockade of the renin angiotensin aldosterone system will provide a substantial benefit through blood pressure lowering independent mechanisms, namely, interruption of fibrogenic pathways, anti-proteinuric actions, amelioration of hyperfiltration and possibly some immunomodulatory effects.

The proposed studies will also characterize the interstitial ultrastructural compositional changes that occur in the renal allografts with CAN, the effects of treatment on these changes and provide a complete description of the incidence and predictors for the development of transplant glomerulopathy. These studies will also determine the impact of angiotensin II receptor blockade on the rate of decline of glomerular filtration rate, as well as the impact of glomerular size on the rate of graft loss from CAN, the incidence and the progression of post transplant proteinuria, the nature of the permselectivity defects responsible for the proteinuria and will also explore the association of proteinuria with graft loss from CAN. This trial will also help construct a profile for the RAAS in the transplant recipients and explore the relationship between two genes polymorphisms, ACE and TGF-Beta, and CAN.

These studies should help to describe the natural history, nature and pathogenesis of CAN, elucidate early markers and predictors of this important disorder and, perhaps, define a safe and useful preventative strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Recipients of a first or a second renal transplant alone or in combination with a pancreas transplantation.
* Informed consent
* Adequate baseline biopsy; at least 10 cortical projection fields.

Exclusion Criteria:

* Age < 18 years.
* Serum creatinine 2.5mg/dL.
* Persistent hyperkalemia; potassium > 5.4 mEq/L.
* Known hypersensitivity to losartan or iodine allergy.
* Documented renal artery stenosis by duplex ultrasonography.
* Recipients of grafts from an HLA-identical sibling.
* Recipients whose primary renal disease is primary hyperoxaluria,dense-deposit disease, focal segmental glomerulosclerosis or hemolytic uremic syndrome.
* Women of childbearing age who wish to become pregnant and/or are unwilling to use contraceptive measures or who are pregnant.
* Recipients requiring ACE inhibitors or AII blockers for a cardiovascular indication (e.g. systolic dysfunction).
* Recipients who are > 55 years old and had a history of cardiovascular disease (coronary artery disease, stroke or peripheral vascular disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2002-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan N. Ibrahim, M.D., M.S., Principal Investigator — University of Minnesota; Bertram Kasiske, M.D., Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (2):
- United States (2):
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data.

REFERENCES:
- [Background] Ibrahim HN, Jackson S, Connaire J, Matas A, Ney A, Najafian B, West A, Lentsch N, Ericksen J, Bodner J, Kasiske B, Mauer M. Angiotensin II blockade in kidney transplant recipients. J Am Soc Nephrol. 2013 Feb;24(2):320-7. doi: 10.1681/ASN.2012080777. Epub 2013 Jan 10. PMID 23308016
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471
- [Derived] Kukla A, Issa N, Jackson S, Spong R, Foster MC, Matas AJ, Mauer MS, Eckfeldt JH, Ibrahim HN. Cystatin C enhances glomerular filtration rate estimating equations in kidney transplant recipients. Am J Nephrol. 2014;39(1):59-65. doi: 10.1159/000357594. Epub 2014 Jan 18. PMID 24457184
- [Derived] Issa N, Ortiz F, Reule SA, Kukla A, Kasiske BL, Mauer M, Jackson S, Matas AJ, Ibrahim HN, Najafian B. The renin-aldosterone axis in kidney transplant recipients and its association with allograft function and structure. Kidney Int. 2014 Feb;85(2):404-15. doi: 10.1038/ki.2013.278. Epub 2013 Aug 21. PMID 23965522

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan: 100 mg/day starting within three months of transplantation
- Placebo: starting within 3 months of transplantation
Period: Overall Study
Arm/Group | Losartan | Placebo
Started | 77 | 76
Completed | 67 | 54
Not Completed | 10 | 22
Not completed — Death | 5 | 7
Not completed — ESRD, Non IF/TA | 1 | 3
Not completed — Withdrawal by Subject | 4 | 12

BASELINE CHARACTERISTICS:
Groups:
- Losartan; Placebo: within 3 months of transplantation
- Total: Total of all reporting groups
Arm/Group | Losartan | Placebo | Total
Number analyzed (Participants) | 77 | 76 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (11.1) | 48.0 (13.6) | 48.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 47 | 47 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 66 | 67 | 133
  Not Available | 11 | 9 | 20
Donor Type [Count of Participants; unit: Participants]
  Live Donor | 53 | 55 | 108
  Cadaver Donor | 24 | 21 | 45
Cause of Native Kidney Disease [Count of Participants; unit: Participants]
  Diabetes mellitus | 28 | 29 | 57
  Hypertension | 8 | 2 | 10
  Polycystic kidney disease | 13 | 10 | 23
  Other | 28 | 35 | 63

OUTCOME MEASURES:

1. Primary Outcome: Doubling of Interstitium or Any ESRD
Description: Doubling of the interstitial or any defined ESRD (including IF/TA)
Time Frame: Baseline to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 48 | 47
Participants | 6 | 12

2. Secondary Outcome: Number of Participants With Cortical Interstitial Volume Expansion or Any ESRD
Description: Number of subjects who had doubling of the interstitial or any end stage renal disease (ESRD) not attributed to interstitial fibrosis and tubular atrophy (IF/TA)
Time Frame: Baseline and 5 Years Post Transplant
Population: Number of subjects who had baseline and exit biopsy samples that could be analyzed for doubling of cortical interstitial volume expansion or graft loss from IF/TA.
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 47 | 44
Participants | 7 | 15

ADVERSE EVENTS:
Time Frame: Subjects were randomized to treatment within three months of organ transplantation and data was collected from baseline to Year 5 post transplantation
Arm/Group | Losartan | Placebo
All-Cause Mortality (participants affected / at risk) | 2/77 | 0/76
Serious Adverse Events (participants affected / at risk) | 77/77 | 76/76
Other Adverse Events (participants affected / at risk) | 35/77 | 42/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Losartan (N=77) | Placebo (N=76)
Bacterial Infection (Infections and infestations) | 15 | 15
Cardiovascular (Cardiac disorders) | 9 | 11
Digestive (Gastrointestinal disorders) | 15 | 18
Endocrine (Endocrine disorders) | 10 | 28
Fungal/Other Infection (Infections and infestations) | 2 | 6
Hematologic (Blood and lymphatic system disorders) | 5 | 10
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 19 | 12
(General disorders) | 14 | 10
Rejection (Immune system disorders) | 12 | 9
Respiratory (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Urogenital (Renal and urinary disorders) | 16 | 26
Viral Infection (Infections and infestations) | 6 | 8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Losartan (N=77) | Placebo (N=76)
Bacterial infection (Infections and infestations) | 4 | 5
Cardiovascular (Cardiac disorders) | 0 | 2
Digestive (Gastrointestinal disorders) | 7 | 4
Endocrine (Endocrine disorders) | 0 | 10
Fungal/other infection (Infections and infestations) | 0 | 2
Hematologic (Blood and lymphatic system disorders) | 2 | 5
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 | 3
Other/Unknown (General disorders) | 3 | 3
Rejection (Immune system disorders) | 5 | 1
Respiratory (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Urogenital (Renal and urinary disorders) | 4 | 5
Viral Infection (Infections and infestations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No